CLINICAL TRIAL: NCT01559597
Title: Etude Comparative de Deux stratégies de Vaccination antitétanique en Situation réelle: Vaccin conservé en chaîne de Froid Versus en chaîne de température contrôlée.
Brief Title: Comparative Study of Two Tetanus Toxoid Vaccination Strategies: Cold Chain Versus Controlled Temperature Chain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Epicentre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Epicentre/CTC-TT/2012
Record Dates: First submitted 2012-03-19; First posted 2012-03-21 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-02

CONDITIONS: Tetanus; Tetanus Vaccine
Keywords: controlled temperature chain; outside the cold chain; vaccination; prevention of mother to child transmission
MeSH Terms: conditions — Tetanus | interventions — Tetanus Toxoid

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Cold chain (Active Comparator): Group vaccinated with tetanus toxoid vaccine kept in cold chain
  Interventions: Biological: Tetanus toxoid vaccine
- CTC (Experimental): Group vaccinated with tetanus toxoid vaccine kept in controlled temperature chain
  Interventions: Biological: Tetanus toxoid vaccine

INTERVENTIONS:
Biological: Tetanus toxoid vaccine — Two doses of tetanus toxoid vaccine separated at least 4 weeks. One arm receives the vaccine kept in cold chain and the other arm receives the vaccine kept in CTC

SUMMARY:
The purpose of this study is to determine the effectiveness, safety and feasibility of a tetanus toxoid (TT) vaccination strategy relying on the maintenance of vaccines in a controlled temperature chain (CTC). The CTC is defined as the storage and transport of vaccines within a temperature range appropriate to the heat stability profile of TT vaccine. In this study vaccines are transported and stored in the cold chain up to district level. From district to beneficiary level vaccines are exposed to ambient temperatures during a limited period of time.

In an initial phase, the stability of 3 lots of TT vaccine kept in CTC is determined. For this, the potency, safety, pH and adsorption of vaccines maintained in CTC will be tested in the laboratory and compared to vaccines that have been maintained in cold chain. If all parameters (i.e. potency, safety, pH and adsorption) are above WHO specifications the strategy in CTC will be used.

Only if the laboratory results are adequate, villages will be assigned to one of the vaccination strategies. All women between 14 to 49 years of age in the selected villages who fulfill the inclusion criteria will be invited to participate.

In order to determine the baseline anti-tetanus protection, TT vaccination history will be collected from all participants using a standardized questionnaire. Women who have already received at least 2 doses of TT vaccine will be excluded from the study. Moreover, blood will be collected from all participants to later verify in laboratory the baseline protection.

A first dose of TT vaccine will be given according to the assigned strategy (CTC or cold chain). Four weeks after the 1st vaccination, a second TT vaccine will be given using the same strategy employed for the first dose. Finally, four weeks after the second dose, a blood sample will be collected from all participants who received two doses of vaccine. The serological responses will be compared in the group that received two doses of TT vaccine maintained in cold chain ant the group that received two doses of vaccine maintained in CTC.

ELIGIBILITY:
Inclusion Criteria:

* Women aged between 14 to 49 years of age
* Living in the district of Moïssala, Chad
* Have no proof of previous vaccination or previous vaccination is not greater than 1 dose of vaccine
* Previous dose received more than 1 month before
* Consented to be included in the study

Exclusion Criteria:

* Allergic reaction to previous tetanus vaccination
* Severe febrile illness
* Have received a tetanus vaccine within the previous month
* Refuses vaccination or does not consent
* Nomadic population travelling before the end of the study
* Pregnant women due to deliver within 2 weeks

Ages: 14 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2129 (Actual)
Dates: Start 2012-11; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Protective level of anti-tetanus antibodies | 4 weeks after second dose of vaccine
  The proportion of women who achieve a protective level of anti-tetanus antibodies after 2 doses of vaccine kept in CTC is not lower to the proportion of women who achieve a protective level of anti-tetanus antibodies after 2 doses of vaccine kept in cold chain.

SECONDARY OUTCOMES:
Vaccine stability | 30 days after exposure to ambient temperatures
  Verify the stability of the vaccine (potency, safety, pH and adsorption) after exposure to ambient temperatures
Antibody levels | 4 weeks after second dose of vaccine
  Evaluate the percentage increase in antibody levels in women who have received 2 doses of vaccine maintained in CTC and in women who have received 2 doses of vaccine maintained in cold chain
Adverse events | 30 min and 7 days after vaccination
  Compare the adverse events in the group vaccinated with the vaccine kept in CTC and the group vaccinated with the vaccine kept in cold chain.

CONTACTS AND LOCATIONS:
Overall Officials: Aitana Juan Giner, MSc, Principal Investigator — Epicentre
Locations (1):
- Moïssala health district, Moïssala, Chad